CLINICAL TRIAL: NCT06893081
Title: An Open-label, Phase 1 Study to Characterize the Effects of a Strong CYP3A4 Inducer on the Pharmacokinetics of MK-8527 in Healthy Adult Participants
Brief Title: A Study of Carbamazepine (CBZ) and MK-8527 in Healthy Adult Participants (MK-8527-012)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 8527-012; MK-8527-012 (Other: MSD)
Record Dates: First submitted 2025-03-18; First posted 2025-03-25 (Actual); Last update posted 2025-07-29 (Actual); Status verified 2025-07

CONDITIONS: Healthy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- MK-8527 + CBZ (Experimental): Treatment A (Period 1): Participants will receive a single dose of MK-8527 on Day 1.
  Treatment B (Period 2): Participants will receive CBZ twice a day on Days 1 to 20 and a single dose of MK-8527 coadministered with the morning dose of CBZ on Day 14.
  A washout period will separate Treatments A and B.
  Interventions: Drug: MK-8527; Drug: CBZ

INTERVENTIONS:
Drug: MK-8527 — Oral Tablet
Drug: CBZ — Oral Extended-release Capsule

SUMMARY:
The goal of this study is to learn what happens to MK-8527 in a healthy person's body over time when MK-8527 is given alone and with the medication CBZ.

ELIGIBILITY:
Inclusion Criteria:

Inclusion criteria include, but are not limited to:

* Is a healthy, adult, male or female of non-childbearing potential only, 18-55 years of age, inclusive
* Is a continuous non-smoker who has not used nicotine- and tobacco-containing products for at least 3 months prior

Exclusion Criteria:

Exclusion criteria include, but are not limited to:

* Has a history or presence of:

  * Seizures (except for febrile seizure), or is at an increased risk for seizures
  * Family history of severe dermatologic reactions including toxic epidermal necrolysis and Stevens-Johnson syndrome
  * Clinically meaningful hematologic diseases, bone marrow disorders, or hematologic adverse reactions to other medications
  * Depression, unusual changes in mood or behavior or suicidal thoughts or behavior
  * Hypersensitivity reaction to anticonvulsant therapy (including phenytoin, primidone, and phenobarbital)
  * Clinically significant eye disease
  * Cardiac conduction disturbance, including second-and third-degree atrioventricular heart block
* Shown to carry or be positive for HLA-A*11:01, HLA-A*31:01, HLA-B*15:02, HLA-B*15:08, HLA-B*15:11, HLA-B*15:21, HLA-B*15:30, or HLA-B*15:31 alleles.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 16 (Actual)
Dates: Start 2025-04-28 (Actual); Primary Completion 2025-06-19 (Actual); Study Completion 2025-07-17 (Actual)

PRIMARY OUTCOMES:
Area Under the Concentration-Time Curve from 0 to Infinity (AUC0-inf) of MK-8527 | Predose and at designated timepoints (up to 168 hours postdose)
  Blood samples will be collected to determine the AUC0-inf of MK-8527 in plasma
Area Under the Concentration-Time Curve from 0 to the Time of the Last Quantifiable Sample (AUC0-last) of MK-8527 | Predose and at designated timepoints (up to 168 hours postdose)
  Blood samples will be collected to determine the AUC0-last of MK-8527 in plasma
Area Under the Concentration-Time Curve from 0 to 24 hours (AUC0-24) of MK-8527 | Predose and at designated timepoints (up to 24 hours postdose)
  Blood samples will be collected to determine the AUC0-24 of MK-8527 in plasma
Area Under the Concentration-Time Curve from 0 to 168 hours (AUC0-168) of MK-8527 | Predose and at designated timepoints (up to 168 hours postdose)
  Blood samples will be collected to determine the AUC0-168 of MK-8527 in plasma
Maximum Observed Plasma Concentration (Cmax) of MK-8527 | Predose and at designated timepoints (up to 168 hours postdose)
  Blood samples will be collected to determine the Cmax of MK-8527 in plasma
Time to Maximum Observed Plasma Concentration (Tmax) of MK-8527 | Predose and at designated timepoints (up to 168 hours postdose)
  Blood samples will be collected to determine the Tmax of MK-8527 in plasma
Apparent Terminal Half-Life (t1/2) of MK-8527 | Predose and at designated timepoints (up to 168 hours postdose)
  Blood samples will be collected to determine the t1/2 of MK-8527 in plasma
Apparent Clearance (CL/F) of MK-8527 | Predose and at designated timepoints (up to 168 hours postdose)
  Blood samples will be collected to determine the CL/F of MK-8527 in plasma
Apparent Volume of Distribution During Terminal Phase (Vz/F) of MK-8527 | Predose and at designated timepoints (up to 168 hours postdose)
  Blood samples will be collected to determine the Vz/F of MK-8527 in plasma

SECONDARY OUTCOMES:
Number of Participants Who Experience an Adverse Event (AE) | Up to approximately 60 days
  An AE is any untoward medical occurrence in a clinical study participant, temporally associated with the use of the study intervention, whether or not considered related to the study intervention.
Number of Participants Who Discontinue Study Treatment Due to an AE | Up to approximately 30 days
  An AE is any untoward medical occurrence in a clinical study participant, temporally associated with the use of the study intervention, whether or not considered related to the study intervention.

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC
Locations (1):
- Celerion ( Site 0001), Tempe, Arizona, United States

IPD SHARING:
Plan to Share IPD: Yes
https://trialstransparency.msdclinicaltrials.com/pdf/ProcedureAccessClinicalTrialData.pdf
URL: https://externaldatasharing-msd.com/

REFERENCES:
- See also: Merck Clinical Trials Information — http://www.merckclinicaltrials.com